CLINICAL TRIAL: NCT07275372
Title: Effectiveness of Virtual Humans in Learning Cognitive Function Assessment Among Nursing Students
Brief Title: Using Virtual Humans to Teach Cognitive Function Assessment to Nursing Students
Acronym: VHCT-NS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N202510056
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Nursing Students

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual human (Experimental): This group will use virtual human to learn the assessement of SPMSQ.
  Interventions: Other: Virtual human
- Printed material (Active Comparator): The comparison group will use printed material to learn the assessment of SPMSQ.
  Interventions: Other: Printed material

INTERVENTIONS:
Other: Virtual human — There are five scenarios integrated into Virtual human software.
  Arms: Virtual human
Other: Printed material — The comparison group will read the printed material regarding SPMSQ assessment.
  Arms: Printed material

SUMMARY:
Purpose of the Study This study wants to find out whether a virtual human (a computer-based simulated person) can help nursing students learn how to assess someone's thinking and memory skills.

Main Question Do nursing students learn cognitive function assessment better when they use a virtual human compared with reading printed materials?

What Participants Will Do Participants will learn how to do a cognitive function assessment for about 60 minutes, either by using a virtual human or by reading printed materials.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students currently enrolled in a bachelor's or post-baccalaureate nursing program.
* Students who have not previously received instruction on the SPMSQ cognitive function assessment,

Exclusion Criteria:

* no

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Competence of cognitive function assessment | 60 minutes
  Participants are required to conduct a cognitive function assessment on the virtual patient within a designed clinical scenario. The system assigns a score based on the completion of each item, with higher scores indicating better cognitive assessment ability.
Knowledge of cognitive function assessment | 60 minutes
  A total of ten items were included. Each correct answer receives one point, while incorrect or "don't know" responses receive zero points. The total score ranges from 0 to 10, with higher scores indicating better knowledge of cognitive function assessment among the students.
Confidence scale | 60 minutes
  The scale consists of five items, each scored from 1 to 5, with a total score ranging from 5 to 25. Higher scores indicate greater confidence in performing cognitive function assessments among the participants.

SECONDARY OUTCOMES:
Learning Material Satisfaction Questionnaire | 60 minutes
  The questionnaire includes 10 items and is scored on a 5-point Likert scale, where "strongly disagree" = 1, "disagree" = 2, "neutral" = 3, "agree" = 4, and "strongly agree" = 5. The total score ranges from 10 to 50, with higher scores indicating greater satisfaction with the learning material (either the VH-based material or the printed material).

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No